CLINICAL TRIAL: NCT02677623
Title: Evaluation of Ureteral Patency in the Post-indigo Carmine Era
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAP3450
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Ureteral Patency
MeSH Terms: interventions — Phenazopyridine; Fluorescein; Mannitol; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A- Pyridium (Experimental): * Method of administration: oral
  * Dose: 200 mg PO with small sip of water
  * Known adverse events: yellow discoloration of skin or sclera, 1-10% central nervous system effects including headache and dizziness, GI effect of cramping, < 1% acute renal failure, methemoglobinemia, hemolytic anemia, hepatitis, rash, skin pigmentation, vertigo, stomach cramps
  * Contraindications: to be used in caution in patients with renal impairment Cr Cl < 50ml/minute and in patients who are receiving nitric oxide, prilocaine and sodium nitrite as it can cause methemoglobinemia
  Interventions: Drug: Pyridium
- B- Sodium Fluorescein (Experimental): * Method of administration: intravenous
  * Dose: 25 mg
  * Known adverse events: nausea, vomiting, flushing or rash, hypersensitivity and anaphylactic reactions can occur following injection and immediate treatment with epinephrine should be available, skin and urine discoloration (urine may appear bright yellow for 24-36 hours), extravasation may cause skin sloughing, toxic neuritis and phlebitis, nausea, rare cardiac arrest and seizure,
  * Contraindications: use with caution in patients with history of hypersensitivity, allergies or asthma
  Interventions: Drug: Sodium Fluorescein
- C- Mannitol (Experimental): * Method of administration: irrigant during cystoscopy
  * Dose: 300cc during cystoscopy to visualize the ureters
  * Known adverse events: dysuria, polyuria, hyponatremia with excess absorption, potential increased risk of urinary tract infection
  * Contraindications when used as a genitourinary irrigation solution: anuria
  Interventions: Drug: Mannitol
- Control- Normal saline (Experimental): * Method of administration: irrigant during cystoscopy
  * Dose: 300cc
  * Known adverse events: no known significant adverse events
  * Contraindications: none
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Pyridium
  Arms: A- Pyridium
Drug: Sodium Fluorescein
  Arms: B- Sodium Fluorescein
Drug: Mannitol
  Arms: C- Mannitol
Other: Normal Saline
  Arms: Control- Normal saline

SUMMARY:
Many gynecologic, urologic and pelvic reconstructive surgeries require accurate ways to identify the opening of the ureters to ensure that they are working correctly. Historically, indigo carmine, an intravenous medication that dyes the urine blue, has been used to help visualize the opening of the ureters with cystoscopy which is a camera placed inside the bladder. In June 2014, the FDA announced there was current shortage of indigo carmine. Thus, investigators need to evaluate other methods for assessing ureteral patency. Ideal alternatives are agents that are low-risk, inexpensive, provide comparable visualization, are readily available and are easy to use.

Examples of such agents currently being used to evaluate the ureters, include oral pyridium, IV sodium fluorescein, and mannitol. These agents help identify the opening of the ureters by either dyeing the urine a different color such as pyridium and sodium fluorescein, or by having a different viscosity to urine such as mannitol. This study will compare three methods of evaluating ureteral patency at time of cystoscopy compared to no method: mannitol, sodium fluorescein, and pyridium.

DETAILED DESCRIPTION:
Many gynecologic, urologic and pelvic reconstructive surgeries require accurate intra-operative evaluation of ureteral patency. Numerous studies show that cystoscopy detects a greater proportion of bladder and ureteral injuries than visual inspection alone.The rate of ureteral injury in gynecologic surgery ranges from 0.6 to 11% when discovered on routine intraoperative cystoscopy depending on the procedure. In a review by Gilmour et al, the incidence of bladder injury in studies performing routine cystoscopy was 4-fold higher than those studies that did not. Early recognition of injury and repair during the primary surgery most often results in less morbidity for the patient, more successful outcome, and increased ease of repair.

Cystourethroscopy is a surgical procedure in which a fiberoptic endoscope is introduced through the urethra to examine the entire lumen of the urethra and bladder for diseases or abnormalities in a systematic manner.There are numerous indications for diagnostic cystourethroscopy during gynecologic surgery. The most important indications are to rule out cystotomy and intravesical or intraurethral suture or mesh placement, verify bilateral ureteral jets to ensure patency, and evaluate a suspected urine leak during or after laparotomy, laparoscopy or vaginal surgery.

Historically, indigo carmine, indigotindisulfonate sodium has been used to assist with cystourethroscopy. Ureteral function is assessed by visualization of ureteral efflux of blue dye after the intravenous injection of indigo carmine. Indigo carmine has many advantages. These include no known drug interactions or metabolites, easy dosing of 40mg or 5 to 10 cc of 0.8% solution, changing urine to a non-physiologic blue color that eases visualization and the ability to give the medication intravenously immediately prior to the procedure. In patients with normal renal function and adequate hydration, the dye is visible after approximately ten minutes, having a half-life of four to five minutes. Because of its large molecular size, it is largely excreted rather than reabsorbed. There are few contraindications to use of indigo carmine. It should be used with caution in patients with cardiovascular diseases secondary to its mild pressor effect.

The U.S. Food and Drug Administration announced the current shortage of indigotindisulfonate sodium in June 2014. This is due to the inability to obtain the active agent. There are two suppliers of indigo carmine in the United States: Akron and American Regent. Akron has discontinued manufacturing indigo carmine with no plan to resume production. American Regent plans to continue manufacturing indigo carmine based on component availability.

Methylene blue is an alternative to indigo carmine. Like indigo carmine, it can be given intravenously. However, it does have some risks. Methylene blue is variably metabolized to multiple end products but is largely metabolized to leukomethylene, which is colorless and therefore, may not be visualized in the urine. It cannot be used in pregnant patients and those with glucose-6-phosphate dehydrogenase deficiency because of risk of inducing hemolytic anemia. It may also cause methemoglobinemia when given in high doses greater than 7mg/kg. Lastly, methylene blue is a monoamine oxidase inhibitor and can cause serotonin syndrome in patients taking other serotonergic agents.

Given the shortage of indigo carmine and the risks associated with use of methylene blue, investigators need to evaluate other methods for assessing ureteral patency. Ideal alternatives are agents that are low-risk, inexpensive, provide comparable visualization, are readily available, and are easy to use. Preoperative oral phenazopyridine and intravenous urelle and sodium fluorescein are other agents that can dye the urine. The use and safety profile of oral phenazopyridine as a bladder analgesic is well established when used for a single short course. Within one hour after ingestion, the urine acquires a characteristic orange tint. A recent study by Hui et al showed that bilateral ureteral patency and bladder mucosal integrity was confirmed in all cases of 124 women that received oral phenazopyridine prior to pelvic surgery. Phenazopyridine is a safe, inexpensive dye that assists effectively in the confirmation of ureteric patency when cystoscopy is planned during pelvic surgery. Consistent with the literature, pyridium has been used at our institution for visualization of the ureters. Some reported concerns include obscuring of the bladder mucosa and a striking similarity between bloody ureteral efflux and pyridium-dyed urine that can be alarming intra-operatively. Doyle et al used sodium fluorescein as an alternative to indigo carmine to assess ureteral patency. This study found that ten percent sodium fluorescein given intravenously in doses ranging from 0.25 to 1.0 cc results in good visualization of ureteral jets. Sodium fluorescein injections have been routinely used for retinal angiography using significantly higher doses than cystoscopy requires. They have proven to be safe and cost effective. A prospective study measuring adverse reactions in patients undergoing ophthalmic angiography found the most common reactions to be nausea (2.9%), vomiting (1.2%) and flushing or rash (0.5%).Mannitol is a low-viscosity, isotonic distending media that is commonly used during hysteroscopy. As the viscosity is different than that of urine, it may allow for better visualization of the flow of urine during cystoscopy. It provides excellent visibility for the endoscopic surgeon but also possesses properties that have a potential impact on patient safety. Five percent mannitol is typically used during transurethral resection or hysteroscopy. Excess mannitol absorption has been known to cause hyponatremia; however, this is an uncommon event. The severity of hyponatremia is directly related to the volume of irrigation fluid that is retained. Absorption greater than 1000mL is typically required to cause clinically significant hyponatremia. In this study, investigators will use only 300mL of mannitol to distend the bladder. Therefore, the risk of hyponatremia is minimal.

ELIGIBILITY:
Inclusion Criteria:

- Planned cystoscopy

Exclusion Criteria:

1. Women who are pregnant
2. Women with contraindications to pyridium, sodium fluorescein or mannitol:

   1. Intra-operative administration of nitric oxide, prilocaine and sodium nitrite
   2. Anuria
   3. Women with creatinine greater than 1 or Cr Cl < 50ml/minute
   4. Known allergy to pyridium, sodium fluorescein or mannitol.
3. Women with a known urologic anatomical anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara Grimes, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 consented subjects were excluded prior to randomization. 8 had completed their surgery during a period of study suspension and 2 ended up not proceeding with surgery.
Groups:
- A- Pyridium: * Method of administration: oral
  * Dose: 200 mg PO with small sip of water
  * Known adverse events: yellow discoloration of skin or sclera, 1-10% central nervous system effects including headache and dizziness, GI effect of cramping, < 1% acute renal failure, methemoglobinemia, hemolytic anemia, hepatitis, rash, skin pigmentation, vertigo, stomach cramps
  * Contraindications: to be used in caution in patients with renal impairment Cr Cl < 50ml/minute and in patients who are receiving nitric oxide, prilocaine and sodium nitrite as it can cause methemoglobinemia
  Pyridium
- B- Sodium Fluorescein: * Method of administration: intravenous
  * Dose: 25 mg
  * Known adverse events: nausea, vomiting, flushing or rash, hypersensitivity and anaphylactic reactions can occur following injection and immediate treatment with epinephrine should be available, skin and urine discoloration (urine may appear bright yellow for 24-36 hours), extravasation may cause skin sloughing, toxic neuritis and phlebitis, nausea, rare cardiac arrest and seizure,
  * Contraindications: use with caution in patients with history of hypersensitivity, allergies or asthma
  Sodium Fluorescein
- C- Mannitol: * Method of administration: irrigant during cystoscopy
  * Dose: 300cc during cystoscopy to visualize the ureters
  * Known adverse events: dysuria, polyuria, hyponatremia with excess absorption, potential increased risk of urinary tract infection
  * Contraindications when used as a genitourinary irrigation solution: anuria
  Mannitol
- Control- Normal Saline: * Method of administration: irrigant during cystoscopy
  * Dose: 300cc
  * Known adverse events: no known significant adverse events
  * Contraindications: none
  Normal Saline
Period: Overall Study
Arm/Group | A- Pyridium | B- Sodium Fluorescein | C- Mannitol | Control- Normal Saline
Started | 33 | 32 | 32 | 33
Completed | 33 | 32 | 32 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A- Pyridium | B- Sodium Fluorescein | C- Mannitol | Control- Normal Saline | Total
Number analyzed (Participants) | 33 | 32 | 32 | 33 | 130
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean age | 52 (11) | 48 (15) | 50 (11) | 52 (12) | NA (NA) — Cannot confirm whether the data was simply not collected for a total mean calculation, or if data was collected but lost. The research team is no longer at Columbia and this information cannot be verified.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 32 | 33 | 130
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4 | 6 | 8 | 4 | 22
  Caucasian | 15 | 7 | 9 | 13 | 44
  Hispanic | 12 | 15 | 13 | 13 | 53
  Asian | 1 | 0 | 1 | 3 | 5
  Other or Unknown | 1 | 4 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: This is a 10-cm visual analog scale to determine which method of evaluating ureteral patency is most satisfactory to physicians. The smiley face is at one end and the frowning face is at the other end. Smiling is 1 and frowning is 10. The scale is completed by surgeon, anesthesiologist and the circulator by placing an "x" or a "mark" anywhere on the 10 cm line towards how good and or bad each person felt about the of process of patency assessment that was used. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from a minimum of 0 to a maximum of 100. A higher score indicates greater pain intensity (worse outcome).
Time Frame: Intraoperative
Population: Inclusion criteria stipulated women age >18 years who desired elective, scheduled gynecologic or urogynecologic surgery. Women were excluded if they were pregnant; had a known urologic anatomical anomaly; or had a history of adverse reaction or contraindication to use of phenazopyridine, sodium fluorescein, or mannitol.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | A- Pyridium | B- Sodium Fluorescein | C- Mannitol | Control- Normal Saline
Number analyzed (Participants) | 33 | 32 | 32 | 33
score on a scale | 48 [0 to 83] | 20 [0 to 82] | 0 [0 to 44] | 28 [3 to 96]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded intraoperatively, 23 hours postoperatively, and at the 2- to 6-week postoperative follow-up visit.
Description: All patient medical records were reviewed for adverse events such as blood transfusion; patient report or provider identification of headache, dizziness, vertigo, stomach cramps, dysuria, polyuria, nausea, vomiting, skin flushing, rash, skin pigmentation, phlebitis, cardiovascular compromise, or skin or sclera discoloration; and abnormal lab values including renal failure ,anemia, and hepatitis , hyponatremia and urinary tract infection (UTI).
Arm/Group | A- Pyridium | B- Sodium Fluorescein | C- Mannitol | Control- Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 2/33 | 1/32 | 1/32 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A- Pyridium (N=33) | B- Sodium Fluorescein (N=32) | C- Mannitol (N=32) | Control- Normal Saline (N=33)
Transfusion (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) — Adverse events within 23 hours of surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No